CLINICAL TRIAL: NCT04832997
Title: Micro-ultrasound or MRI-targeted Biopsy for Prostate Cancer Diagnosis
Brief Title: Micro-ultrasound for Prostate Cancer Diagnosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study faced structural and methodological obstacles, with limited enrollment, technical issues, low adherence, and loss of scientific relevance.
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Alberto Briganti, Full Professor, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: US-MIRROR
Record Dates: First submitted 2021-04-03; First posted 2021-04-06 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Every patient will receive the same diagnostic test (MRI and Micro-US) in a randomized sequence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mpMRI plus Micro-US (Experimental): Patients with a clinical suspicion of csPCa will receive mpMRI and Micro-US in two different visits (randomized sequence). The results of the diagnostic procedures will determine how many and which type of prostate biopsies patients will undergo.
  Interventions: Diagnostic Test: Prostate biopsy systematic random prostate biopsy (TRUS-Bx) + eventual MRI-targeted biopsy (MRI-TBx) + eventual microUS-targeted (Micro-US-TBx)

INTERVENTIONS:
Diagnostic Test: Prostate biopsy systematic random prostate biopsy (TRUS-Bx) + eventual MRI-targeted biopsy (MRI-TBx) + eventual microUS-targeted (Micro-US-TBx) — Patients with both positive mpMRI and Micro-US, defined as the presence of one or more lesions with PI-RADS >= 3 and PRI-MUS >= 3 respectively, will receive a 12-core TRUSBx in addiction to MRI-TBx and Micro-US-TBx. Patients with both negative mpMRI and Micro-US will receive a 12-core TRUSBx. Patients with only positive mpMRI will receive MRI-TBx and 12-core TRUSBx. Patients with only positive Micro-US-TBx will receive Micro-US-TBx and 12-core TRUSBx.

SUMMARY:
This is a single-center, paired-cohort, prospective study. Patients with a clinical suspicion of csPCa will receive mpMRI and Micro-US in two different visits. The results of the diagnostic procedures will determine how many and which type prostate biopsies patients will undergo. During the following visit, patients with both positive mpMRI and Micro-US, defined as the presence of one or more lesions with PI-RADS ≥ 3 and PRI-MUS ≥ 3 respectively, will receive a 12-core TRUSBx in addiction to MRI-TBx and Micro-US-TBx (Group 4). Patients with both negative mpMRI and Micro-US will receive a 12-core TRUSBx (Group 1). Patients with only positive mpMRI will receive MRI-TBx and 12-core TRUSBx (Group 2). Patients with only positive Micro-US-TBx will receive Micro-US-TBx and 12-core TRUSBx (Group 3).

Our hypothesis is that the sensitivity for csPCa (defined as prostate cancer with Gleason score ≥ 3+4) of Micro-US will be superior or at least equal to that of mpMRI. Despite the introduction of the mpMRI and MRI-TBx has improved the diagnostic pathway of PCa, the proportion of men with negative mpMRI with a csPCa is still difficult to delineate due to the high variability of mpMRI negative predictive value (NPV) and specificity. In this context, a specific standardization of the use of Micro-US may play a crucial role to optimize PCa diagnostic pathway. Moreover, a direct comparison between Micro-US and mpMRI might be useful to determinate whether Micro-US could be more accurate than mpMRI for PCa diagnosis. Furthermore, in patients with suspicion of PCa the combined use between mpMRI and Micro-US might increase the detection of csPCa and reduce the number of unnecessary biopsies, improving mpMRI limitations in NPV and specificity. Demonstrating that Micro-US provides a similar sensitivity for csPCa as compared to mpMRI may lead to its definitive inclusion in daily clinical practice, potentially replacing mpMRI, streamlining the current diagnostic pathway of PCa.

ELIGIBILITY:
Inclusion Criteria:

* Men at least 18 years of age referred with clinical suspicion of prostate cancer who have been advised to have a prostate biopsy
* Serum PSA ≤ 20ng/ml
* Suspected stage ≤ T2 on rectal examination (organ-confined prostate cancer)
* Fit to undergo all procedures listed in protocol
* Able to provide written informed consent

Exclusion Criteria:

* Prior treatment for prostate cancer
* Prior diagnosis of prostate cancer
* Contraindication to MRI (e.g. claustrophobia, pacemaker, estimated GFR ≤ 50mls/min)
* Contraindication to prostate biopsy
* Men in whom artifact would reduce the quality of the MRI
* Previous hip replacement surgery, metallic hip replacement or extensive pelvic orthopaedic metal work
* Unfit to undergo any procedures listed in protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Sensitivity in detecting clinically significant prostate cancer of Micro-US vs. mpMRI | through study completation, an average time of 2 years
  To compare the sensitivity in detecting clinically significant prostate cancer of Micro-US vs. mpMRI

SECONDARY OUTCOMES:
Proportion of clinically significant prostate cancer detected with the inclusion of Micro-US within the diagnostic pathway of prostate cancer | through study completation, an average time of 2 years
  To report the diagnostic benefit related with the use of Micro-US in the prostate cancer diagnostic pathway
Proportion of men with clinically insignificant prostate cancer detected by MRI-TBx vs. Micro-US-TBx | through study completation, an average time of 2 years
Proportion of men with at least one lesion detected by mpMRI vs. Micro-US | through study completation, an average time of 2 years
Proportion of men with clinically significant prostate cancer detected by Micro-US-TBx missed by MRI-TBx and vice-versa | through study completation, an average time of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy